CLINICAL TRIAL: NCT01950624
Title: DS-Connect®: The Down Syndrome Registry
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Linda Crnic Institute for Down Syndrome (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-0396; OT2HD117033 (NIH)
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Down Syndrome
Keywords: Patient Registry; Down Syndrome; Natural History
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Down syndrome cohort: Individuals who have a diagnosis of complete trisomy 21, translocation Down syndrome or mosaic Down syndrome.

SUMMARY:
The goal of this study is to develop a registry for Down syndrome (DS) to facilitate research participation by individuals with Down syndrome.

DS-Connect® is an online survey tool designed to collect demographic data and health information from individuals with DS. It is open to all people with Down syndrome.

The purposes of DS-Connect® are:

1. To identify the various phenotypic manifestations of DS.
2. To identify individuals with DS who may be eligible for research studies or new clinical trials, based on specific information about their diagnosis and health history.

DETAILED DESCRIPTION:
The DS-Connect® Registry is a unique resource that enables communication and sharing of ideas among the NIH, individuals with DS and their families, national and international organizations interested in DS, and a diverse group of professionals involved in scientific research and medical care benefiting the population with DS. By providing information on their demographics, health histories, medications, and other relevant biomedical information, self-advocates and their families provide an unprecedented view of this genetic condition that can inspire new scientific inquiries, clinical research, and clinical trials specifically serving this population. For example, the DS-Connect® dataset has led to an increasing appreciation of the prevalence of many co-occurring conditions affecting individuals with DS across the lifespan, thus providing the rationale for the launch of the NIH INCLUDE Project (INvestigation of Co-occurring conditions across the Lifespan to Understand Down SyndromE). Conversely, self-advocates and their families participating in DS-Connect® benefit in several ways, including valuable comparison of their health histories with metrics from the entire cohort, access to key resources (e.g., list of active clinical trials), as well as opportunities for participation in human research protocols, including clinical trials testing new interventions to address diverse aspects of this condition. In turn, the DS-Connect® dataset informs both NIH and the research community on the need to support specific research areas, while also providing an avenue for researchers to promote recruitment into their studies. Altogether, DS-Connect® provides a multimodal platform for exchange of information and ideas across all key stakeholders, assuring that scientific research in this field is attuned to the needs of the community.

A person with DS or a family member or caregiver can register directly through the DS-Connect® website at their convenience. They may learn of the Registry from many sources including partner advocacy groups, government and healthcare organizations, or other families who are members in the Registry. The DS-Connect® platform readily captures participant information using condition-specific surveys.

All information is provided by the participant or representative for the participant via the web-based Registry. There are no in-person visits required for registration.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adults (at least 18 years of age) with a diagnosis of DS (including mosaic DS or partial trisomy 21) who are capable of providing consent to participate, or for whom a legally authorized representative (LAR) may give permission on behalf of the individual to participate. Adults with DS who cannot consent for themselves but can provide assent would need to provide assent to their LAR.
* Children (up to age 18 years of age) with a diagnosis of DS. Parents/guardians may enter registry information and give permission to participate on behalf of their child; if the child is over 7 years of age and able to provide assent, they must do so. (Note: Once a child has reached age 18, he or she will be prompted to re-enroll into the registry as an adult, if he/she is able to provide informed consent or with the consent of his/her LAR if unable to re-enroll themselves.)

No individuals with DS will be excluded from taking part in DS-Connect based on age, race, ethnicity, or gender.

EXCLUSION CRITERIA:

* A person who does not have a diagnosis of DS (or mosaic DS or partial trisomy 21)
* Adults with DS who are not capable of providing informed consent or assent to participate and do not have a Legally Authorized Representative who can do so. In the case where an adults with DS is able to provide assent but does not do so, that adult will be excluded.
* A participant, parent, and/or LAR who cannot provide consent or does not read or understand a language that is available for the registry, either English or Spanish.
* A child with DS (between the ages of 7 and 18 years) who is capable of providing assent but does not do so.
* A child under the age of 18 years whose parents share joint custody and one parent indicates that they do not consent to the child's participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with DS (including those with mosaic DS and partial trisomy 21).
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2013-09-06 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
To determine the prevalence of the various co-occurring conditions in Down syndrome. | Through study completion, up to 10 years
  Participants in DS-Connect® will complete health history surveys regarding medical diagnoses and can update the surveys annually or whenever their health changes.
Facilitate participation in research for individuals with DS who may be eligible for research studies or new clinical trials. | Through study completion, up to 10 years
  Participants may choose to hear about Down syndrome research studies that may be relevant to their co-occurring conditions.

SECONDARY OUTCOMES:
Enable aggregate data sharing from individuals with Down syndrome. | Through study completion, up to 10 years
  Consented individuals will have their de-identified data shared with the INCLUDE Data Hub to enable researchers to understand etiology, natural history, and/or treatment effectiveness in Down syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin M Espinosa, Ph.D., Principal Investigator — Linda Crnic Institute for Down Syndrome, University of Colorado Anschutz Medical Campus
Locations (1):
- Linda Crnic Institute for Down Syndrome, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other researchers through the INCLUDE Data Hub.